CLINICAL TRIAL: NCT06282341
Title: Fatigue and Recovery: a Comparison Between Trail and Marathon
Acronym: MARA-TRAIL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 23CH132
Record Dates: First submitted 2023-10-23; First posted 2024-02-28 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: Running; Marathon; Trail; Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: Prospective study on healthy volunteers, comparing the neurophysiological, physiological and biomechanical effects at the end of a marathon compared with an equivalent effort trail in the open air, or simulated on a treadmill, in runners specialising in each of the 2 disciplines
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MARASIM (Active Comparator): During visit 2, road runners will take part in a simulated marathon race on a treadmill.
  Interventions: Other: Race: Simulated marathon
- TRAILSIM (Active Comparator): During visit 2, trail runners will take part in a simulated trail race on a treadmill.
  Interventions: Other: Race: Simulated trail
- TRAILNAT (Active Comparator): During visit 2, trail runners will take part in a real trail race in the nature.
  Interventions: Other: Race: Trail in nature

INTERVENTIONS:
Other: Race: Simulated marathon — Participants will take part in a race: simulated marathon. Before, during, immediately after and the month after the race, neuromuscular, physiological and biomechanical assessments will take place.
  Arms: MARASIM
Other: Race: Simulated trail — Participants will take part in a race: simulated trail. Before, during, immediately after and the month after the race, neuromuscular, physiological and biomechanical assessments will take place.
  Arms: TRAILSIM
Other: Race: Trail in nature — Participants will take part in a race: trail in nature. Before, during, immediately after and the month after the race, neuromuscular, physiological and biomechanical assessments will take place.
  Arms: TRAILNAT

SUMMARY:
Road marathon is a famous running race known for hundreds of years. Trail running is an emerging running discipline which count new runners every year. Trail running and road marathon are two running endurance disciplines which differed by variation of elevation and nature of the terrain. While marathon is essentially run on flat roads, trail races are realized on steep paths (mountain, desert…) with an important variation of elevation. Neuromuscular, biomechanical and physiological consequences are different depending on the discipline, especially with a greater eccentric contribution in trail running. In spite of this characteristic, trail runners take part in several races longer than 40 km per year, while road runners participate in one to two marathons per year.

DETAILED DESCRIPTION:
Some studies focused on fatigue and recovery following 30-to-40-km trail races or marathon but no direct comparison between both disciplines have been done yet. A direct comparison between marathon and trail would aim to better understand if the occurrence of fatigue is more important or if the recovery is longer in one of the two disciplines. The comparison is also a way to better understand mechanisms involved in fatigue and recovery following a trail and a marathon. Then, this research could be applied to improve specificity of training and prevent risk of injuries. This project aims to compare fatigue and recovery following a trail and a marathon.

ELIGIBILITY:
Inclusion Criteria:

Common for MARASIM, TRAILSIM and TRAILNAT:

* Male or female
* 18-55 years old
* Endurance runners who run at least one running session of 20 km per week
* Being able to run a marathon under 5 h or finishing a trail of 30 km during the last 3 years
* Refrain from participating to a competition one month before the first visit and during the duration of the study
* To have a medical certificate of no contraindication of running practise in competition
* Registered with a social security scheme
* Having given the written consent freely

Specific for the 3 groups :

* Specialist of trail running (TRAILSIM and TRAILNAT)
* Specialist of road running (MARASIM)

Exclusion Criteria:

* Subjects who present cardiac or articular chronic pathologies (example: repeated sprain, patellar or joint problems)
* Subjects who present chronic or central neurological pathologies
* Subjects deprived of liberty or who should be legally deprived
* Subjects who report to take forbidden products by the World Anti-Doping Agency
* pregnant or breastfeeding woman

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-12-28 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in knee extensors maximal isometric torque output | Day 0 (day of the race) baseline value = 30 minutes before the race and 15 minutes after the race
  The primary outcome will be changed (in % of baseline value) of the maximal voluntary torque (in Nm) produced by the knee extensors, measured at D0 (= day of the race) with an isometric knee dynamometer (ARS dynamometry, SP2, Ltd., Ljubljana, Slovenia), before (baseline value = 30 minutes before the race) and at the end (15 minutes after the race) of a marathon or a trail (depending on the group)

SECONDARY OUTCOMES:
Change in plantar flexor maximal isometric torque output | Day 0 (day of the race) baseline value = 30 minutes before the race and 15 minutes after the race, Days 1, 2, 7
  Change (in % of baseline value) of the maximal voluntary torque (in Nm) produced by the plantar flexor measured at D0, by an instrumental pedal placed at 45 degrees with respect to the horizontal (ATI Industrial Automation, Inc., Apex, North Carolina USA), before (baseline value) and at the end of a marathon or a trail (depending on the group), and during recovery at Day1 Day2 Day7).
Recovery of quadriceps maximal isometric torque output the month after the race | Day 0 (day of the race) baseline value = 30 minutes before the race, (Day 1 (= 24 hours after the end of the race) , Day 2 (= 48 hours after the end of the race), Day 7 (= 7 days after the end of the race).
  Change (in % of post-exercise baseline value) of the maximal voluntary torque (in Nm) produced by the knee extensors, measured with an isometric knee dynamometer (ARS dynamometry, SP2, Ltd., Ljubljana, Slovenia), during recovery at Day 1 Day 2 Day 7).
Voluntary activation level | D0 (day of the race) baseline value = 30 min before the race, in the middle of the race (except for the trail in the nature) and 15 min after the race;D1 = 24h after the end of the race , D2 = 48h after the end of the race, D7 = 7 days after the end
  Voluntary activation level (in %) of the plantar flexors and knee extensors will be assessed through neuromuscular assessments before, in the middle (except for the trail in the nature), after the marathon or trail of equivalent effort, and during recovery (Day 1, Day 2, and Day 7).
  Voluntary activation level will be calculated as followed:
  VA (%) = (1- (superimposed Db100/ resting Db100))x100
Force assessed in dynamic | Day 0 15 minutes before the race, after the marathon or trail ( 1 hour after the end), and during recovery (Day 1 (= 24 hours after the end of the race) , Day 2 (= 48 hours after the end of the race), Day 7 (= 7 days after the end of the race).
  Force assessed in dynamic mode on a cycloergometer (Monark, Vansbro, Sweden) composed of strain gauges, a flywheel, a belt and an optical encoder allowing data collection. Force (N) will be measured in order to establish a force-velocity / power- velocity profile at Day 0 15 min before the race, after the marathon or trail ( 1 hour after the end) of equivalent effort, and during recovery (Day 1 (= 24h after the end of the race) , Day 2 (= 48 h after the end of the race), Day 7 (= 7 days after the end of the race).
Velocity assessed in dynamic | Day 0 15 minutes before the race, after the marathon or trail ( 1 hour after the end), and during recovery (Day 1 (= 24 hours after the end of the race) , Day 2 (= 48 hours after the end of the race), Day 7 (= 7 days after the end of the race).
  Velocity assessed in dynamic mode on a cycloergometer (Monark, Vansbro, Sweden) composed of strain gauges, a flywheel, a belt and an optical encoder allowing data collection. Speed (rad/s) will be measured in order to establish a force-velocity / power-velocity profile before (=15 minutes before the race), after the marathon or trail (=1 hour after the end) of equivalent effort, and during recovery (Day 1 = 24hours after the end of the race, Day 2 = 48hours after the end of the race, Day 7 = 7 days after the end of the race).
Power assessed in dynamic | Day 0 15 minutes before the race, after the marathon or trail ( 1 hour after the end), and during recovery (Day 1 (= 24 hours after the end of the race) , Day 2 (= 48 hours after the end of the race), Day 7 (= 7 days after the end of the race).
  Power assessed in dynamic mode on a cycloergometer (Monark, Vansbro, Sweden) composed of strain gauges, a flywheel, a belt and an optical encoder allowing data collection. Power (W) will be measured in order to establish a force-velocity / power-velocity profile before (=15 minutes before the race), after the marathon or trail (=1 hour after the end) of equivalent effort, and during recovery (Day 1 = 24hours after the enf of the race, Day 2 = 45hours after the end of the race, Day 7= 7 days after the race).
Muscular power and stretch-shortening cycle assessed through squat jumps | Day 0 15 minutes before the race, after the marathon or trail ( 1 hour after the end), and during recovery (Day 1 (= 24 hours after the end of the race) , Day 2 (= 48 hours after the end of the race), Day 7 (= 7 days after the end of the race).
  Muscular power and stretch-shortening cycle assessed through squat jump ; Height (m) and duration (s) of jumps are calculated through force platform (90 x90 cm, Model 9287C, Kisler, Winterthur, Switzerland).
Muscular power and stretch-shortening cycle assessed through countermovement jump | Day 0 15 minutes before the race, after the marathon or trail ( 1 hour after the end), and during recovery (Day1 (= 24 hours after the end of the race) , Day 2 (= 48 hours after the end of the race), Day 7 (= 7 days after the end of the race).
  Muscular power and stretch-shortening cycle assessed through countermovement. Height (meter) and duration (seconde) of jumps are calculated through force platform (90 x90 centimeter, Model 9287C, Kisler, Winterthur, Switzerland)
Muscular power and stretch-shortening cycle assessed through drop jump | Day 0 15 minutes before the race, after the marathon or trail ( 1 hour after the end), and during recovery (Day 1 (= 24hours after the end of the race) , Day 2 (= 48 hours after the end of the race), Day 7 (= 7 days after the end of the race).
  Muscular power and stretch-shortening cycle assessed through drop jump. Height (m) and duration (s) of jumps are calculated through force platform (90 x90 cm, Model 9287C, Kisler, Winterthur, Switzerland)
Muscle electrical activity | Day 0: 30 minutes before the race, in the middle (except for the trail in the nature) 15 minutes after the end of the race
  Muscle electrical activity (Trigno avanti Sensor, Delsys, Natick, MA including electrodes connected to thin-10-cm-long cables) are measured
The kinetics of energy cost | Day 0 1 hour 30 minutes before the race,in the middle, 30 minutes after the end of the race, and during recovery (Day 1 (= 24hours after the end of the race) , Day 2 (= 48 hours after the end of the race), Day 7 (= 7 days after the end of the race).
  The kinetics of energy cost (Ccr en J/kg/m) measured using a portable gas exchange measurement system (Ergospirometer Metamax 3B®, Cortex Medical, Leipzig, Germany) 1h30 before the race, in the middle (except for the trail in the nature) and 30 min after the race the marathon or simulated trail and during recovery Day 1, Day 2, Day 7 7)7).measurement system (Ergospirometer Metamax 3B®, Cortex Medical, Leipzig, Germany)
Racing kinematics | 1 hour before, in the middle and immediately after the race and during recovery(Day 1 (= 24hours after the end of the race) , Day 2 (= 48 hours after the end of the race), Day 7 (= 7 days after the end of the race).
  Evolution of moments and hip joint angles, knee and ankle measured by a Markerless tracking system will be measured
  1 hour before the race , in the middle (except for the trail in the nature), immediately after the simulated trail or marathon, and during recovery (Day 1 (= 24hours after the end of the race) , Day 2 (= 48hours after the end of the race), Day 7 (= 7 days after the end of the race).
Ground reaction force (in Newton) | 1hour before, in the middle (except for the trail in the nature) and immediately after the race and during recovery(Day 1 (= 24hours after the end of the race) , Day 2 (= 48hours after the end of the race), Day 7 (= 7 days after the end of the race).
  Force will be measured by force platforms contained in the treadmill (h/p/Cosmos-Stellar, Germany). to get the ground reaction forces at each step 1hour before, in the middle (except for the trail in the nature) and immediately after the race and during recovery(Day 1 (= 24hours after the end of the race) , Day 2 (= 48hours after the end of the race), Day 7 (= 7 days after the end of the race).
Center of pressure (in Newton) | 1hour before, in the middle (except for the trail in the nature) and immediately after the race and during recovery(Day 1 (= 24hours after the end of the race) , Day 2 (= 48 hours after the end of the race), Day 7 (= 7 days after the end of the race).
  Force will be measured by force platforms contained in the treadmill (h/p/Cosmos-Stellar, Germany). to get the center of pressure each step before (=1 hour before), in the middle (except for the trail in the nature), after (=immediately after the race) the simulated trail or marathon, and during recovery (Day 1 = 24 hours after the race, Day 2 = 48 hours after the race, Day 7 = 7 days after the race)
Muscle damage blood markers | Day 0: 2hours before the race, 2hours after the race and during recovery (Day 1 (= 24hours after the end of the race) , Day 2 (= 48 hours after the end of the race), Day 7 (= 7 days after the end of the race).
  Witness muscle damage following a marathon or a trail of equivalent effort. Biological variables are taken 2h before the race and 2 h after the race: a marathon or a trail of equivalent effort, and during recovery ((Day 1 (= 24h after the end of the race) , Day 2 (= 48 hours after the end of the race), Day 7 (= 7 days after the end of the race). Followed i- Inflammatory parameters are taken through blood test (2 tubes of 5 ml/blood test): ionogram (sodium [mmol/l], potassium [mmol/l], chlorine [mmol/l], bicarbonates [mmol/l], urea [mmol/l], creatinine [µmol/l], glucose [mmol/l], proteins [g/l], uric acid [[µmol/l ], osmolality [m0smol/kg]; Creatine Kinase (UI/l)myoglobine [µg/l ], C reactive Protein [mg/l], lactate [mmol/l]
Resting heart rate variability parameters | 3 times in the 2 weeks before the race and every other day for the month following the race
  Evolution of resting heart rate variability, a marker of psychophysiological recovery will be assessed through a Polar H10 heart rate monitor before the race (at least 3 times in the 2 weeks before the race) and during recovery (at least every two days until one month after the race).
  Analysis of time domain and frequency domain variables via measurement of heart rate variability will be achieved through HRV analysis software.
Effort perception | D0 (day of the race) : during the race, every 5 kilometers effort
  Perception of effort will be assessed during the marathon or trail of equivalent effort every 5 km effort on the modified Borg scale (from 0 - rest to 10 - Maximal perceived effort).
Fatigue assessment | Once during 2 weeks before, immediately after the race and during recovery (Day 1 = 24 hours after the race, Day 2 = 48 hours after, Day 3 = 72 hours after, Day 4, Day 5, Day 6, Day 7, Day 14, Day 21 and Day 30 after the race
  Fatigue assessment will be carried out before (=once during the 2 weeks before the race) the marathon or trail of equivalent effort , immediately after and during recovery (Day 1 = 24 hours after the race, Day 2 = 48 hours after the race, Day 3 = 72 hours after the race, Day 4 = 4 days after the race, Day 5 = 5 days after the race, Day 6 = 6 days after the race, Day 7 = 7 days after the race, Day 14 = 14 days after the race, Day 21 = 21 days after the race, Day 30 = 30 days after the race) via the of the "Rating scale of fatigue " (from 0 - Not fatigued at all to 10 - Total exhaustion nothing left).
Muscular pain | Day 0 (day of the race) : during the race, every 5 kilometers effort
  Muscle pain felt in the quadriceps and calves will be rated on a visual analog scale ranging from 0 (No muscular pain at all) at 10 (Unbearable muscle pain) during the marathon or trail of equivalent effort every 5 km-effort

CONTACTS AND LOCATIONS:
Overall Officials: Leonard FEASSON, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Unités de Myologie et de Médecine du Sport, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No